CLINICAL TRIAL: NCT01262196
Title: A Multi-center, Randomized, Double-blind, Controlled Study to Evaluate the Safety and Efficacy of MP4OX Treatment, in Addition to Standard Treatment, in Severely Injured Trauma Patients With Lactic Acidosis Due to Hemorrhagic Shock
Brief Title: Phase IIb Study of MP4OX in Traumatic Hemorrhagic Shock Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sangart (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TRA-205
Record Dates: First submitted 2010-12-15; First posted 2010-12-17 (Estimated); Last update posted 2013-08-22 (Estimated); Status verified 2013-08

CONDITIONS: Shock, Hemorrhagic; Shock, Traumatic; Acidosis, Lactic
Keywords: Trauma; Hemorrhage; Hemorrhagic shock; Lactic acidosis; Oxygen carriers; Oxygen therapeutics; Hemoglobin solutions; Red cell substitutes; PEG-hemoglobin
MeSH Terms: conditions — Shock, Hemorrhagic; Shock, Traumatic; Acidosis, Lactic; Wounds and Injuries; Hemorrhage | interventions — polynitroxylated pegylated hemoglobin; maleimide-polyethylene glycol-modified hemoglobin, MP4; PEG-hemoglobin; Sodium Chloride; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MP4OX (Experimental): 250-mL dose
  Interventions: Drug: MP4OX
- Control (Placebo Comparator): 250-mL of normal saline solution
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: MP4OX — 4.3 g/dL pegylated hemoglobin in balanced lactate-electrolyte solution
  Other Names: Hemoglobin pegylated; MalPEG-Hb; MP4; PEG-Hb; Pegylated-Hb
  Arms: MP4OX
Drug: Saline — Normal saline (0.9%) solution
  Other Names: Normal saline; Saline solution; Sodium chloride 0.9%
  Arms: Control

SUMMARY:
MP4OX is a novel oxygen therapeutic agent being developed as an ischemic rescue therapy to enhance perfusion and oxygenation of tissues at risk during hemorrhagic shock. MP4OX is a pegylated hemoglobin-based colloid. Due to its molecular size and unique oxygen dissociation characteristics, MP4OX targets delivery of oxygen to ischemic tissues. This study will evaluate the safety and efficacy of MP4OX treatment in trauma patients suffering from lactic acidosis due to severe hemorrhagic shock. The study hypothesis is that MP4OX will reverse the lactic acidosis by enhancing perfusion and oxygenation of ischemic tissues and thereby prevent and reduce the duration of organ failure and improve outcome in these patients.

DETAILED DESCRIPTION:
Acute traumatic injury, including both blunt and penetrating injury, is often associated with severe uncontrolled bleeding which can lead to hemorrhagic shock. During shock, inadequate blood flow results in local ischemia and tissue hypoxia (insufficient oxygenation) of critical organs, which can be detected by an increase in serum lactate levels in these trauma victims. Despite optimal care, more than 10% of trauma victims who reach hospital alive will die, and many will suffer from organ failure. Death and significant, persistent morbidity are consequences of trauma, and traumatic injuries are associated with lost productivity, reduced quality of life, and direct costs to patients and health care systems worldwide.

The primary treatment of trauma is to support ventilation and oxygenation, limit blood loss, and maintain cardiovascular function so that organs are perfused. The patient's airway may be intubated to allow oxygenated airflow to the lungs. Mechanical ventilation is used if the patient cannot maintain oxygenation and carbon dioxide elimination. Damage-control surgery is used to limit blood loss and to intentionally delay definitive repair until the patient can better tolerate procedures. Blood transfusions are provided to maintain the oxygen-carrying capacity of the circulation. Platelets and coagulation factors are infused to correct any coagulopathy from dilution of blood and consumption of clotting factors. Vasopressor and inotropic agents may be used to support low cardiac output or blood pressure. Renal replacement therapy may be instituted if kidney failure occurs.

Despite optimal care, organ dysfunction is present in many patients. Hypoperfusion and anaerobic metabolism of organs and tissues can be detected by the presence of lactic acidosis. Current therapy is aimed at supporting failing organs, but an agent that accelerates the repayment of an oxygen debt and prevents or shortens the duration of organ failure is sought. Blood transfusion improves circulation of oxygen-carrying red blood cells but is insufficient if lactic acidosis is present, even when the hemoglobin level has been restored. Studies in critically ill intensive care patients have demonstrated that elevated initial and 24-hour lactate levels are significantly correlated with mortality, and prolonged elevation of blood lactate levels after trauma has been correlated with increased organ failure and mortality.

Support for the efficacy of MP4OX in resuscitation of severe hemorrhage shock comes from several preclinical studies in hamster, rat, and swine. Using a swine model of uncontrolled hemorrhage and resuscitation, survival was greater and restoration of hemodynamics and acid-base status were improved with MP4OX relative to equivalent volume of crystalloid, pentastarch, or unmodified hemoglobin. Administration of MP4OX improved 24-hour survival, stabilized cardiac output and arterial pressure at nearly normal levels, and reduced lactate more effectively than control fluids. Importantly, these benefits of MP4OX were observed with or without co-administration of autologous blood, suggesting that blood alone is not sufficient to achieve resuscitation, and that the effects of MP4OX are additional to those of blood.

Additional support comes from a recently completed phase IIa trauma study in 51 patients with lactic acidosis due to severe hemorrhage. MP4OX treatment was associated with a more rapid and sustained reduction of high lactate levels, and a greater proportion of MP4OX-treated patients who normalized lactate by four hours after dosing. There was also a trend toward shorter median hospital stay and a greater proportion of MP4OX-treated patients being discharged from hospital alive by Day 28. These phase IIa results suggest improved oxygen delivery and utilization by ischemic tissues in the MP4OX-treated patients, based on the reversal of lactic acidosis, and support the positive results from the preclinical models of hemorrhagic shock resuscitation.

ELIGIBILITY:
Inclusion Criteria:

* Adult male or female (surgically sterile or post-menopausal or confirmed not to be pregnant)
* Trauma injury (blunt and/or penetrating) resulting in lactic acidosis due to hemorrhagic shock
* Acidosis (blood lactate level ≥ 5 mmol/L; equivalent to 45 mg/dL) arterial or venous

Exclusion Criteria:

* Massive injury incompatible with life
* Normalization of lactate prior to dosing (≤ 2.2 mmol/L)
* Patients with evidence of severe traumatic brain injury as defined by ANY one of the following: Known non-survivable head injury or open brain injury; Glasgow Coma Score (GCS) = 3, 4 or 5; Known AIS (head region) ≥ 4 shown by an appropriate imaging methodology; Contemplated CNS surgery; or Abnormal physical exam indicative of severe CNS or any spinal cord injury above T5 level
* Cardiac arrest prior to randomization
* Age below the legal age for consenting
* Estimated time from injury to randomization> 4 hours
* Estimated time from hospital admission to randomization > 2 hours
* Known pregnancy
* Use of any oxygen carrier other than RBCs
* Known previous participation in this study
* Professional or ancillary personnel involved with this study
* Known receipt of any investigational drug(s) within 30 days prior to study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 348 (Actual)
Dates: Start 2011-05; Primary Completion 2012-10 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Proportion of patients discharged from hospital through day 28 and alive at the Day 28 follow-up visit | 28 days

SECONDARY OUTCOMES:
Hospital-free, ICU-free, and ventilator-free days | Through 28 days
Composite endpoint of Time to Complete Organ Failure Resolution (CTCOFR) | At 14 and 21 days
Proportion of patients who normalize (≤ 2.2 mmol/L) lactate levels | 2, 4, 6, 8 and 12 hours
Proportion of patients remaining: (1) in hospital, (2) in ICU, and (3) on ventilator through Day 28 | 28 days
Number of days: (1) in hospital, (2) in ICU, and (3) on the ventilator | Through 28 days
All-cause mortality | At 48 hours and at 28 days
Time (days) from randomization to: (1) death, (2) discharge from hospital, (3) discharge from ICU, and (4) liberation from mechanical ventilation | Through 28 days
Sequential organ failure assessment (SOFA score) | Daily
Modified Denver score | Daily

CONTACTS AND LOCATIONS:
Overall Officials: Karim Brohi, MD, Principal Investigator — The Royal London Hospital
Locations (40):
- Australia (2):
  - Liverpoool Hospital NSW, Liverpool
  - John Hunter Hospital, Newcastle
- Graz University Hospital, Gratz, Austria
- Brazil (3):
  - Faculdade de Medicina de S. J. Do Rio Preto, São José do Rio Preto
  - Hospital das Clínicas - USP, São Paulo
  - Hospital Universitário - USP Ribeirão Preto, São Paulo
- Fundacion Valle de Lili, Cali, Colombia
- France (8):
  - Hôpital Beaujon, Clichy
  - Hôpital Michallon, Grenoble
  - Hôpital du Kremlin Bicêtre, Le Kremlin-Bicêtre
  - Hôpital Roger Salengro, CHRU Lille, Lille
  - Hôpital Dupuytren, CHU Limoges, Limoges
  - Hôpital Edouard Herriot, Lyon
  - Hôpital Lyon sud, Lyon
  - Hôpital Pitié-Salpêtrière, Paris
- Germany (5):
  - Universitätsklinikum der RWTH Aachen, Aachen
  - Charite - Campus Virchow Klinikum, Berlin
  - Kliniken der Stadt Köln Merheim, Cologne
  - Klinikum der Johann-Wolfgang-Goethe-Universität Frankfurt a.M., Frankfurt
  - BG Klinik Ludwigshafen, Ludwigshafen
- Israel (3):
  - Soroka University Medical Center, Beersheba
  - Rambam Hospital, Haifa
  - Hadassah Medical Center, Jerusalem
- Auckland Hospital, Auckland, New Zealand
- Oslo university hospital, Oslo, Norway
- Singapore (3):
  - National University Hospital, Singapore
  - Singapore General Hospital, Singapore
  - Tan Tock Seng Hospital, Singapore
- South Africa (6):
  - Netcare Union Hospital, Alberton
  - Vincent Pallotti Hospital, Cape Town
  - Netcare Unitas Hospital, Centurion
  - Charlotte Maxeke Johannesburg Hospital, Johannesburg
  - Netcare Milpark Hospital, Johannesburg
  - Chris Baragwanath Hospital, Soweto
- Hospital 12 de Octubre, Madrid, Madrid, Spain
- Switzerland (2):
  - Centre Hospitalier Universitaire Vaudois CHUV, Lausanne
  - Universitätsspital Zürich, Zurich
- United Kingdom (3):
  - King's College Hospital, London, London
  - The Royal London Hospital, London
  - John Radcliffe Hospital, Oxford, Oxford

REFERENCES:
- [Background] Young MA, Lohman J, Malavalli A, Vandegriff KD, Winslow RM. Hemospan improves outcome in a model of perioperative hemodilution and blood loss in the rat: comparison with hydroxyethyl starch. J Cardiothorac Vasc Anesth. 2009 Jun;23(3):339-47. doi: 10.1053/j.jvca.2008.08.006. Epub 2008 Oct 22. PMID 18948027
- [Background] Young MA, Riddez L, Kjellstrom BT, Winslow RM. Effect of maleimide-polyethylene glycol hemoglobin (MP4) on hemodynamics and acid-base status after uncontrolled hemorrhage in anesthetized swine: comparison with crystalloid and blood. J Trauma. 2007 Dec;63(6):1234-44. doi: 10.1097/TA.0b013e31815bd7b0. PMID 18212644
- [Background] Young MA, Riddez L, Kjellstrom BT, Bursell J, Winslow F, Lohman J, Winslow RM. MalPEG-hemoglobin (MP4) improves hemodynamics, acid-base status, and survival after uncontrolled hemorrhage in anesthetized swine. Crit Care Med. 2005 Aug;33(8):1794-804. doi: 10.1097/01.ccm.0000172648.55309.13. PMID 16096458
- [Background] Drobin D, Kjellstrom BT, Malm E, Malavalli A, Lohman J, Vandegriff KD, Young MA, Winslow RM. Hemodynamic response and oxygen transport in pigs resuscitated with maleimide-polyethylene glycol-modified hemoglobin (MP4). J Appl Physiol (1985). 2004 May;96(5):1843-53. doi: 10.1152/japplphysiol.00530.2003. Epub 2004 Jan 16. PMID 14729723
- [Background] Vandegriff KD, Winslow RM. Hemospan: design principles for a new class of oxygen therapeutic. Artif Organs. 2009 Feb;33(2):133-8. doi: 10.1111/j.1525-1594.2008.00697.x. PMID 19178457
- [Background] Vandegriff KD, Malavalli A, Mkrtchyan GM, Spann SN, Baker DA, Winslow RM. Sites of modification of hemospan, a poly(ethylene glycol)-modified human hemoglobin for use as an oxygen therapeutic. Bioconjug Chem. 2008 Nov 19;19(11):2163-70. doi: 10.1021/bc8002666. PMID 18837531
- [Background] Svergun DI, Ekstrom F, Vandegriff KD, Malavalli A, Baker DA, Nilsson C, Winslow RM. Solution structure of poly(ethylene) glycol-conjugated hemoglobin revealed by small-angle X-ray scattering: implications for a new oxygen therapeutic. Biophys J. 2008 Jan 1;94(1):173-81. doi: 10.1529/biophysj.107.114314. Epub 2007 Sep 7. PMID 17827244
- [Background] Winslow RM, Lohman J, Malavalli A, Vandegriff KD. Comparison of PEG-modified albumin and hemoglobin in extreme hemodilution in the rat. J Appl Physiol (1985). 2004 Oct;97(4):1527-34. doi: 10.1152/japplphysiol.00404.2004. Epub 2004 Jun 18. PMID 15208289
- [Background] Tsai AG, Cabrales P, Manjula BN, Acharya SA, Winslow RM, Intaglietta M. Dissociation of local nitric oxide concentration and vasoconstriction in the presence of cell-free hemoglobin oxygen carriers. Blood. 2006 Nov 15;108(10):3603-10. doi: 10.1182/blood-2006-02-005272. Epub 2006 Jul 20. PMID 16857991
- [Background] Tsai AG, Vandegriff KD, Intaglietta M, Winslow RM. Targeted O2 delivery by low-P50 hemoglobin: a new basis for O2 therapeutics. Am J Physiol Heart Circ Physiol. 2003 Oct;285(4):H1411-9. doi: 10.1152/ajpheart.00307.2003. Epub 2003 Jun 12. PMID 12805024
- [Background] Olofsson CI, Gorecki AZ, Dirksen R, Kofranek I, Majewski JA, Mazurkiewicz T, Jahoda D, Fagrell B, Keipert PE, Hardiman YJ, Levy H; Study 6084 Clinical Investigators. Evaluation of MP4OX for prevention of perioperative hypotension in patients undergoing primary hip arthroplasty with spinal anesthesia: a randomized, double-blind, multicenter study. Anesthesiology. 2011 May;114(5):1048-63. doi: 10.1097/ALN.0b013e318215e198. PMID 21455059
- [Background] van der Linden P, Gazdzik TS, Jahoda D, Heylen RJ, Skowronski JC, Pellar D, Kofranek I, Gorecki AZ, Fagrell B, Keipert PE, Hardiman YJ, Levy H; 6090 Study Investigators. A double-blind, randomized, multicenter study of MP4OX for treatment of perioperative hypotension in patients undergoing primary hip arthroplasty under spinal anesthesia. Anesth Analg. 2011 Apr;112(4):759-73. doi: 10.1213/ANE.0b013e31820c7b5f. Epub 2011 Feb 11. PMID 21317165
- See also: Sangart Inc. (San Diego, CA) web site — http://www.sangart.com